CLINICAL TRIAL: NCT01682759
Title: A Phase III, Multicenter, Double-Blind, Randomized Study to Evaluate the Safety and Efficacy of the Addition of MK-3102 Compared With the Addition of Glimepiride in Subjects With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin
Brief Title: A Study of the Safety and Efficacy of Omarigliptin (MK-3102) Compared With Glimepiride in Participants With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin (MK-3102-016)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3102-016; MK-3102-016 (Other: protocol number)
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; glimepiride; Metformin; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omarigliptin (Experimental): Participants will receive omarigliptin, 25 mg once weekly and placebo matching glimepiride once daily for up to 54 weeks.
  Interventions: Drug: Omarigliptin; Drug: Glimepiride Placebo; Drug: Metformin; Drug: Insulin Glargine
- Glimepiride (Active Comparator): Participants will receive glimepiride titrated to a maximum of 6 mg, once daily, and placebo to omarigliptin, once weekly for up to 54 weeks.
  Interventions: Drug: Placebo to Omarigliptin; Drug: Glimepiride; Drug: Metformin; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Omarigliptin
  Arms: Omarigliptin
Drug: Placebo to Omarigliptin
  Arms: Glimepiride
Drug: Glimepiride — Glimepiride (1 mg and/or 2 mg tablets). During the 54-week double-blind treatment period, glimepiride can be up-titrated, as appropriate, to a maximum total daily dose of 6 mg/day. Throughout the trial, down-titration of glimepiride may also occur based upon the participant's glucose measurements and clinical symptoms of hypoglycemia.
  Other Names: AMARYL®; GLIMY
  Arms: Glimepiride
Drug: Glimepiride Placebo
  Arms: Omarigliptin
Drug: Metformin — Participants will continue on their stable dose (>=1500 mg/day) of open-label metformin throughout the trial.
Drug: Insulin Glargine — Insulin glargine can be used for rescue therapy, if glycemic control is not maintained. Insulin therapy should be initiated as per local country insulin glargine label.

SUMMARY:
This trial will assess the safety and efficacy of omarigliptin (MK-3102) compared with the sulfonylurea, glimepiride, in Type 2 diabetes mellitus participants with inadequate glycemic control on metformin monotherapy. The primay hypothesis of the study is that after 54 weeks, the mean change from baseline in hemoglobin A1C (A1C) in participants treated with omarigliptin is non-inferior compared with that in participants treated with glimepiride.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 diabetes mellitus
* On a stable dose of metformin (≥1500 mg/day) for at least 12 weeks with inadequate glycemic control
* Females of reproductive potential agree to remain abstinent or use or have their partner use acceptable methods of birth control

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* Treated with any antihyperglycemic agents (AHA) therapies other than the protocol-required metformin within the prior 12 weeks of study participation or with omarigliptin at any time prior to signing informed consent
* On a weight loss program and is not in the maintenance phase or has

started a weight loss medication in the past 6 months or has undergone bariatric surgery within 12 months prior to study participation

* Medical history of active liver disease (other than non-alcoholic

hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease

* Human immunodeficiency virus
* New or worsening coronary heart disease, congestive heart failure, myocardial infarction, unstable angina, coronary artery intervention, stroke or transient ischemic neurological disorder within the past 3 months
* History of malignancy ≤5 years prior to study participation except for adequately treated basal cell or squamous cell skin cancer, or in situ

cervical cancer

* Clinically important hematological disorder (such as aplastic anemia,

myeloproliferative or myelodysplastic syndromes, thrombocytopenia)

* Pregnant or breast-feeding, or is expecting to conceive or donate eggs

during the trial, including 21 days following the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2012-09-10 (Actual); Primary Completion 2015-01-26 (Actual); Study Completion 2015-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Handelsman Y, Lauring B, Gantz I, Iredale C, O'Neill EA, Wei Z, Suryawanshi S, Kaufman KD, Engel SS, Lai E. A randomized, double-blind, non-inferiority trial evaluating the efficacy and safety of omarigliptin, a once-weekly DPP-4 inhibitor, or glimepiride in patients with type 2 diabetes inadequately controlled on metformin monotherapy. Curr Med Res Opin. 2017 Oct;33(10):1861-1868. doi: 10.1080/03007995.2017.1335638. Epub 2017 Jun 28. PMID 28548024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 1197 participants at 115 clinical sites were screened and 446 participants were excluded during screening. The most common reason for participants not being randomized was screen failure. The most common reasons for screen failure were participants not meeting the metformin inclusion criteria or meeting exclusionary laboratory values.
Period: Overall Study
Arm/Group | Omarigliptin | Glimepiride
Started | 376 | 375
Treated | 375 | 375
Completed | 307 | 305
Not Completed | 69 | 70
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 10 | 13
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 56 | 55

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omarigliptin | Glimepiride | Total
Number analyzed (Participants) | 376 | 375 | 751
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (9.6) | 57.6 (9.3) | 57.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 164 | 337
  Male | 203 | 211 | 414
Hemoglobin A1C [Mean (Standard Deviation); unit: A1C (%)] — For both the Omarigliptin and Glimepiride groups n=375
  A1C (%) | 7.49 (0.75) | 7.43 (0.72) | 7.46 (0.73)
Fasting Plamsa Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — For both the Omarigliptin and Glimepiride groups n=375
  mg/dL | 155.3 (31.4) | 152.7 (30.0) | 154.0 (30.7)
Body Weight [Mean (Standard Deviation); unit: kg] — For both the Omarigliptin and Glimepiride groups n=375
  kg | 87.5 (18.1) | 88.7 (18.7) | 88.1 (18.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C at Week 54
Description: Hemoglobin A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). Thus, this change from baseline reflects the Week 54 A1C minus the Week 0 A1C.
Time Frame: Baseline and Week 54
Population: The Full Analysis Set (FAS) population consisted of all randomized participants who received at least 1 dose of study medication and had a baseline measurement or a measurement for the analysis endpoint after receiving study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C (%)
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 375 | 375
A1C (%) | -0.30 [-0.39 to -0.21] | -0.48 [-0.57 to -0.39]
Statistical Analysis 1: Comparison: Omarigliptin vs Glimepiride; Test type: Non-Inferiority or Equivalence — Omarigliptin was considered non-inferior to glimepiride if the upper bound of the two-sided 95% confidence interval (CI) of the between-treatment difference in least-squares (LS) means for change from baseline in A1C at Week 54 (omarigliptin vs. glimepiride) was lower than 0.35%; Difference in the least squares means = 0.18, 95% CI 2-sided [0.06 to 0.30] — Constrained longitudinal data analysis (cLDA) model including terms for treatment, time, and the interaction of time by treatment, with the constraint that the mean baseline is the same for all treatment groups

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event Excluding Data After Glycemic Rescue
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Time Frame: Up to Week 57
Population: All Subjects as Treated (ASaT) population, defined as all randomized participants who received at least 1 dose of study medication. Participants were included in the treatment group corresponding to the study treatment they actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 375 | 375
Percentage of participants | 54.7 | 61.6
Statistical Analysis 1: Comparison: Omarigliptin vs Glimepiride; Test type: Superiority or Other; Difference in percentages = -6.9, 95% CI 2-sided [-13.9 to 0.1] — Miettinen & Nurminen method; the 95% CI was computed only for those endpoints with at least 4 participants having events in one or more treatment groups

3. Primary Outcome: Percentage of Participants Who Discontinued From the Study Due to an Adverse Event Excluding Data After Glycemic Rescue
Time Frame: Up to Week 54
Population: The ASaT Population is defined as all randomized participants who received at least 1 dose of study medication. Participants were included in the treatment group corresponding to the study treatment they actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 375 | 375
Percentage of participants | 3.7 | 2.7
Statistical Analysis 1: Comparison: Omarigliptin vs Glimepiride; Test type: Superiority or Other; Difference in percentages = 1.1, 95% CI 2-sided [-1.6 to 3.8] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 54
Description: Blood glucose was measured on a fasting basis. FPG is expressed as mg/dL. Blood was drawn at predose on Day 1 and after 54 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 54 minus FPG at baseline).
Time Frame: Baseline and Week 54
Population: The FAS population consisted of all randomized participants who received at least 1 dose of study medication and had a baseline measurement or a measurement for the analysis endpoint after receiving study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 375 | 375
mg/dL | -2.7 [-6.7 to 1.3] | -8.3 [-12.4 to -4.3]
Statistical Analysis 1: Comparison: Omarigliptin vs Glimepiride; Test type: Superiority or Other; Difference in the least squares means = 5.6, 95% CI 2-sided [0.1 to 11.2] — cLDA model including terms for treatment, time, and the interaction of time by treatment, with the constraint that the mean baseline is the same for all treatment groups

5. Secondary Outcome: Percentage of Participants Achieving a Hemoglobin A1C of <6.5% at Week 54
Description: The percentage of participants who achieved A1C values <6.5% (48 mmol/mol) in the FAS Population at Week 54.
Time Frame: Week 54
Population: The FAS Population (with multiple imputation) consisted of all randomized participants who received at least 1 dose of study medication and had a baseline measurement or a measurement for the analysis endpoint after receiving study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 375 | 375
Percentage of participants | 25.1 [20.6 to 30.2] | 28.8 [24.1 to 34.0]
Statistical Analysis 1: Comparison: Omarigliptin vs Glimepiride; A1C <6.5%; Test type: Superiority or Other; Between-group Rate Difference (%) = -3.7, 95% CI 2-sided [-10.6 to 3.3] — Between-group CIs are calculated via Miettinen & Nurminen method

6. Secondary Outcome: Percentage of Participants With an Adverse Event of Symptomatic Hypoglycemia Excluding Data After Glycemic Rescue
Description: Symptomatic episode of hypoglycemia was an episode with clinical symptoms reported by the investigator as hypoglycemia (concurrent fingerstick glucose not required).
Time Frame: Up to Week 54
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 375 | 375
Percentage of participants | 5.3 | 26.7
Statistical Analysis 1: Comparison: Omarigliptin vs Glimepiride; Test type: Superiority or Other; p < 0.001, Difference in percentages; Difference in percentages = -21.3, 95% CI 2-sided [-26.5 to -16.4] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Change From Baseline in Body Weight at Week 54 Excluding Data After Gylcemic Rescue
Time Frame: Baseline and Week 54
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 375 | 375
kg | -0.4 [-0.8 to -0.0] | 1.5 [1.1 to 1.9]
Statistical Analysis 1: Comparison: Omarigliptin vs Glimepiride; Test type: Superiority or Other; p < 0.001, Difference in the least squares means; Difference in the least squares means = -1.9, 95% CI 2-sided [-2.5 to -1.4] — cLDA model including terms for treatment, time, and the interaction of time by treatment with the constraint that the mean baseline is the same for all treatment groups

8. Secondary Outcome: Percentage of Participants Achieving a Hemoglobin A1C of <7.0% at Week 54
Description: The percentage of participants who achieved A1C values <7.0% (53 mmol/mol) in the FAS Population at Week 54.
Time Frame: Week 54
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 375 | 375
Percentage of participants | 47.7 [42.3 to 53.1] | 58.0 [52.7 to 63.1]
Statistical Analysis 1: Comparison: Omarigliptin vs Glimepiride; A1C < 7.0%; Test type: Superiority or Other; Between-group Rate Difference = -10.3, 95% CI 2-sided [-17.8 to -2.8] — Between-group CIs are calculated via Miettinen & Nurminen method

ADVERSE EVENTS:
Time Frame: Up to Week 57
Description: Serious adverse events are presented, regardless of time from last dose of blinded study medication, including data after glycemic rescue. Non-serious adverse events are presented, regardless of time from last dose of blinded study medication, excluding data after glycemic rescue.
Arm/Group | Omarigliptin | Glimepiride
Serious Adverse Events (participants affected / at risk) | 24/375 | 18/375
Other Adverse Events (participants affected / at risk) | 43/375 | 125/375
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (N=375) | Glimepiride (N=375)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic arthritis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Dumping syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (N=375) | Glimepiride (N=375)
Nasopharyngitis (Infections and infestations) | 24 (31) | 23 (30)
Hypoglycaemia (Metabolism and nutrition disorders) | 21 (45) | 110 (487)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.